CLINICAL TRIAL: NCT02025504
Title: Efficacy of ColoWrap® Abdominal Binder in Improving Performance and Tolerance of Colonoscopy: a Randomized, Sham-Controlled, Blinded Clinical Trial
Brief Title: Carolina-ColoWrap® in Colonoscopy Performance and Outcomes Study
Acronym: C3PO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ColoWrap, LLC (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ColoWrap-002
Record Dates: First submitted 2013-12-28; First posted 2014-01-01 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Performance and Tolerance of Colonoscopy
Keywords: Colonoscopy, Looping, Sigmoid Looping, ColoWrap, Binder, Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ColoWrap Intervention Group (Experimental): Patients randomized to ColoWrap Intervention Group will have the ColoWrap abdominal binder secured firmly around their lower abdomen just prior to colonoscopy.
  Interventions: Device: ColoWrap
- Sham Group (Sham Comparator): Sham Group will also have a ColoWrap binder placed around their lower abdomen, but it will be placed loosely so no appreciable lower abdominal pressure is generated by the device.
  Interventions: Device: ColoWrap

INTERVENTIONS:
Device: ColoWrap — ColoWrap is an abdominal binder intended as an accessory to facilitate colonoscopy.
  Other Names: ColoWrap abdominal binder; ColoWrap colonoscopy binder; ColoWrap device; ColoWrap binder

SUMMARY:
Colonoscopy is the gold-standard for colorectal cancer screening in the US. However, complete colonoscopy can be a challenging technical procedure, even for expert gastroenterologists due to variations in patient anatomy, tortuous colons, and looping of the endoscope. Such obstacles can prolong colonoscopy, lead to complications, decrease polyp detection, and impact patient experience and tolerance. The investigators propose to evaluate the efficacy of a new non-invasive abdominal binder (ColoWrap®) in improving the performance and tolerance of colonoscopy by way of a randomized, blinded clinical trial. Eligible participants undergoing colonoscopy at University of North Carolina Hospitals (UNCH) will be recruited for the study and randomized to either the ColoWrap intervention or sham arm. Colonoscopy will be performed per usual operating procedures. The primary outcome will be time to distal extent (cecal intubation time). Secondary outcomes include colonoscopy completion rate, use of ancillary maneuvers, medication usage, procedural difficulty, patient comfort, and operator and assistant fatigue and pain. Efficacy will be assessed on the basis of pairwise comparisons between groups with respect to primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults between the ages of 40 - 80
* Undergoing a colonoscopy at any of the study locations for:

  i. CRC screening (first colonoscopy or 10 year follow up of negative exam). ii. Surveillance (prior colonoscopy with polyps). iii. Diagnostic colonoscopy performed to evaluate symptoms such as abdominal pain or rectal bleeding.
* Participants must have completed the full prescribed colonoscopy purgative preparation prior to their procedure, and describe adequate cleansing.
* For the purposes of informed consent, participants must be able to understand and read English.

Exclusion Criteria:

* Inability to provide informed consent
* Active or suspected pregnancy
* Patients referred due to incomplete colonoscopy or for removal of difficult polyps
* History of problems with sedation or anesthesia -. Participants electing to be unsedated for colonoscopy
* Patients undergoing multiple procedures (e.g. upper and lower endoscopy)
* Previous colon resection surgery
* Patients with known or suspected diagnosis of inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* Patients with a history of colorectal cancer or other intra-abdominal malignancy.
* Patients with open or recent wounds or skin rash on the anterior abdominal wall.
* History of cirrhosis or ascites
* Known ventral or umbilical hernia
* Patients who are medically unstable(American Society of Anesthesiology Class III or above).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean colonoscopic insertion time | During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified
  Colonoscopic insertion time will be defined as the time from insertion of the colonoscope into the rectum to identification of the base of the cecum

SECONDARY OUTCOMES:
Frequency of use of ancillary maneuvers | During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified
  Binary data indicating individually whether abdominal pressure or patient position change was used during the insertion phase of the procedure will be recorded.
Frequency of prolonged, difficult cases | During colonoscopy, from time point of insertion of scope into rectum to point in time when scope is removed from rectum
  The frequency of prolonged, difficult cases. Procedures in which the insertion phase is greater than 20 min will be recorded and indicated as such.
Drug and Dosage Required to Complete Procedure | During colonoscopy, from time point of insertion of scope into rectum to point in time when scope is removed from rectum
  Drug and dosage amount required by patient to complete colonoscopy.
Colonoscopy Completion Rate | During colonoscopy, from time point of insertion of scope into rectum to point in time when scope is removed from rectum
  Colonoscopy completion rate. Dichotomous outcome indicating if the procedure was incomplete or complete.
Time to patient discharge | From time point in which scope is removed from patient's rectum following a colonoscopy until the time the patient is discharged from the facility
  Time to discharge, defined as the time from withdrawal of the colonoscope to patient discharge from the endoscopy unit.
Operator perception of patient discomfort | During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified
  Immediately following completion of procedure, ColoWrap study assistant will obtain operator perception of patient discomfort during procedure according to the Gloucester score
Patient Pain, Bloating, and Satisfaction at Discharge | At single time point occurring after the colonoscopy, just prior to the patient being discharged from facility
  The ColoWrap study assistant will interview patient just prior to discharge and obtain responses for pain and bloating according to 10-point visual analog scales, and global satisfaction according to a 5-point scale.
Operator's Assessment of Procedural Difficultly | During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified
  Immediately following completion of procedure, the study assistant will obtain the operator's assessment of procedural difficulty and level of physical fatigue according to 5-point scales.
Assistant/Technician's Assessment of Musculoskeletal Pain Following Procedure | During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified
  The study assistant will ask the endoscopy technician if they experienced pain during the procedure in any of the following four anatomical sites: lower back, upper back, neck, or upper extremities (right and left shoulder, arm, wrist, hand, fingers). This frequency data will be dichotomous.

OTHER OUTCOMES:
Patient Assessment of Intra-Procedural Pain | During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified
  For patients undergoing colonoscopy with conscious sedation, the study assistant will also obtain a response for intra-procedural pain, using a validated measure of procedural comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Seth D Crockett, MD, MPH, Principal Investigator — Division of Gastroenterology and Hepatology, University of North Carolina, Chapel Hill, NC
Locations (3):
- United States (3):
  - UNC Hospitals, Chapel Hill, North Carolina
  - UNC Meadowmont Endoscopy Center, Chapel Hill, North Carolina
  - UNC Hillsborough Endoscopy Center, Hillsborough, North Carolina

REFERENCES:
- [Derived] Crockett S, Dellon ES, Biggers L, Ernst DA. Use of Patient Abdominal Compression Device Reduces Staff Musculoskeletal Pain Associated With Supporting Colonoscopy: Results From a Randomized Controlled Trial. Gastroenterol Nurs. 2021 Mar-Apr 01;44(2):136-145. doi: 10.1097/SGA.0000000000000550. PMID 33795622
- [Derived] Crockett SD, Cirri HO, Kelapure R, Galanko JA, Martin CF, Dellon ES. Use of an Abdominal Compression Device in Colonoscopy: A Randomized, Sham-Controlled Trial. Clin Gastroenterol Hepatol. 2016 Jun;14(6):850-857.e3. doi: 10.1016/j.cgh.2015.12.039. Epub 2016 Jan 6. PMID 26767313